CLINICAL TRIAL: NCT02822352
Title: A Comparison Of High Definition White Light And High Definition Virtual Chromoendoscopy For The Detection Of Intraepithelial Neoplasia In Longstanding Colitis: A Randomised Controlled Trial
Brief Title: RCT: HDWL vs Virtual Chromoendoscopy in the Detection of Intraepithelial Neoplasia in Longstanding Colitis
Acronym: VIRTUOSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHT/2016/02
Record Dates: First submitted 2016-06-29; First posted 2016-07-04 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis; Crohn's Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Definition White Light (No Intervention): Surveillance colonoscopy using High Definition White Light alone
- High Definition Virtualchromoendoscopy (Active Comparator): High Definition Virtualchromoendoscopy
  Interventions: Other: Chromoendoscopy

INTERVENTIONS:
Other: Chromoendoscopy — High definition virtual chromoendoscopy
  Arms: High Definition Virtualchromoendoscopy

SUMMARY:
Colitis is inflammation of the large bowel and it is often caused by conditions known as ulcerative colitis and Crohn's disease. In these conditions, the body has an exaggerated inflammatory response against the bowel - the body attacks the bowel. Patients who have had colitis affecting most of the large bowel for more than 8 years are at increased risk of cancer of the large bowel. In view of this, many national gastroenterology organisations have recommended that such patients have regular colonoscopies to detect pre-cancerous areas and even early cancer in the large bowel. Early detection of such areas, will lead to early treatment thereby reducing the risk of developing significant large bowel cancer. These regular colonoscopies are known as surveillance colonoscopies.

Official international guidelines for surveillance in patients with ulcerative and Crohn's colitis advise to take 4 random samples of large bowel tissue (biopsies) every 10 centimeters and of any suspicious areas. Recent studies have shown that spraying dye such as indigo carmine (a type of food dye) helps highlight abnormal areas that could harbor pre-cancerous cells. This technique is time-consuming, and tedious. There are no set standards of what is considered a satisfactorily completed dye spray colonoscopy. The uptake of this technique in the UK has not been uniform. Therefore virtual chromoendoscopy has been studied as an alternative method to improve the detection of pre-cancerous tissue in patients with longstanding colitis.

DETAILED DESCRIPTION:
Virtual chromoendoscopy systems enhances specific characteristics of the lining of the large bowel such as surface patterns and mucosal vasculature. This theoretically increases the detection of pre-cancerous tissue compared to high definition white light endoscopy alone. Narrow-band imaging or NBI (Olympus, Tokyo, Japan), Blue Laser (Fujinon, Tokyo, Japan) and OE scan (Pentax, Tokyo, Japan) use optical light filters to select particular narrow spectrums of red, green and blue light with a relative decrease in the proportion of red light. The Fujinon Intelligent Chromo-Endoscopy (FICE) system uses post hoc computer algorithms, applying different filters to the stored endoscopic images and enabling a theoretically endless number of combinations of filters that can be used. The Pentax I-SCAN system also allows post hoc modification of the images. It provides the ability to enhance the mucosal surface to better highlight mucosal changes.

These new imaging techniques have a theoretical advantage, which is extendedly used for sales purposes but so far has not been proven in the surveillance for precancerous or early cancer of the large bowel in patients with longstanding colitis.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative Colitis or Crohn's colitis with a disease duration of >8 years for pancolitis or >15 years duration for left-sided colitis
* Aged 18 years and above
* Patients able to give informed consent

Exclusion Criteria:

* Persistent coagulopathy or platelet count <50x1012 which may preclude mucosal biopsy
* Known colonic IN or CRC
* Fulminant colitis
* Patients who have been previously randomised and withdrawn on 2 occasions due to poor bowel preparation
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-08; Primary Completion 2018-03-08 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
To compare the rates of neoplasia detection using virtual chromoendoscopy compared to high definition white light (HDWL) endoscopy | 14 months

SECONDARY OUTCOMES:
To assess the neoplasia detection rate in targeted biopsies versus non-targeted (segmental) biopsies within each arm of the study | 14 months
  The above is assessed by comparing the mean neoplasia per patient detection rate between virtual chromoendoscopy and high definition white light endoscopy as well as by assessing the yield of non-targeted quadratic biopsies in detecting neoplasia
To compare the duration of time taken using each technique | 14 months
  This is measured by assessing the total withdrawal time taken in each arm of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandiah K, Subramaniam S, Thayalasekaran S, Chedgy FJ, Longcroft-Wheaton G, Fogg C, Brown JF, Smith SC, Iacucci M, Bhandari P. Multicentre randomised controlled trial on virtual chromoendoscopy in the detection of neoplasia during colitis surveillance high-definition colonoscopy (the VIRTUOSO trial). Gut. 2021 Sep;70(9):1684-1690. doi: 10.1136/gutjnl-2020-320980. Epub 2020 Nov 19. PMID 33214162